CLINICAL TRIAL: NCT05762822
Title: Exogenous Ketone Ester in Women with Polycystic Ovary Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1-10-72-217-22
Record Dates: First submitted 2023-02-15; First posted 2023-03-10 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: PCOS
Keywords: 3-hydroxybutyrate; ketones; metabolism; testosterone; androgens; KetoneAid; Ketone monoester
MeSH Terms: conditions — Ketosis | interventions — Water

STUDY DESIGN:
Intervention Model Description: Power calculation resulted in n=18 for the primary endpoint. We plan to include n= 20 to ensure statistical power and take dropouts, missing values etc into account.
  Washout period of minimum 3 days.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 60 ml water (same taste as active comparator) at 10 pm the night before and 6 am on the day for blood sampling (8 am).
  Interventions: Dietary Supplement: water
- 3-OHB (Active Comparator): 60 ml 3-OHB (30 g) at 10 pm the night before and 6 am on the day for blood sampling (8 am).
  Interventions: Dietary Supplement: 3-OHB (KE4)

INTERVENTIONS:
Dietary Supplement: 3-OHB (KE4) — 60 ml (30 g) of 3-OHB
  Other Names: ketone supplement
  Arms: 3-OHB
Dietary Supplement: water — 60 ml water (added bitter taste)
  Arms: Placebo

SUMMARY:
Polycystic ovarian syndrome (PCOS) is characterized by elevated androgens such as testosterone. Clinical studies suggest that ketogenic diets lower the levels of androgens. The ketone 3-hydroxybutyrate (3-OHB) may play an important role in these effects and the main purpose of this study is to investigate whether a 3-OHB supplement acutely improves the hormonal and metabolic status in women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 5-18% of women and is characterized by the presence of two of three of the Rotterdam criteria: Hyperandrogenism (clinical or biochemical), irregular menstrual cycles, and polycystic ovary morphology, after exclusion of other conditions that mimic PCOS. PCOS is associated with elevated levels of luteinizing hormone (LH) and unaltered levels of the follicle stimulating hormone (FSH), which leads to the characteristic hyperandrogenism (high levels of testosterone), oligo- or anovulation, and a large number of premature follicles in the ovarian. Insulin resistance causes hyperinsulinemia that decreases sex hormone binding globulin (SHBG) levels and stimulates androgen production (e.g., elevated concentrations of testosterone). Ketogenic diets are characterized by a diet low in carbohydrates, and has shown beneficial effects on weight and hormonal status in women with PCOS. Whether these improvements are mediated by ketones (e.g., 3-hydroxybutyrate, 3-OHB) or other effects related to this diet is unknown. The main purpose of this study is to investigate whether a 3-OHB supplement acutely improves the hormonal and metabolic status in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnosis
* age >18 years

Exclusion Criteria:

* Medications affecting sex hormones (e.g. contraceptives, dopamine agonists, etc) or glucose metabolism (e.g. saxenda).
* Anemia (Hgb < 6.0 mM)
* Practicing ketogenic diets (e.g., low-carb diet, fasting regimes)
* Inability to understand Danish or English
* Diabetes
* Ongoing cancer or other acute/chronic serious diseases (PI will determine)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of testosterone | 10 hours after first intervention
  Paired t-test

SECONDARY OUTCOMES:
plasma SHBG | 10 hours after first intervention
plasma 3-OHB | 10 hours after first intervention
plasma glucose | 10 hours after first intervention
serum insulin | 10 hours after first intervention
plasma C-peptide | 10 hours after first intervention
plasma free fatty acids | 10 hours after first intervention
plasma triglycerides | 10 hours after first intervention
plasma cholesterol | 10 hours after first intervention
C reactive protein | 10 hours after first intervention
plasma cytokines (such as Tumor Necrotic Factor alpha, Interleukin 6, Lipopolysaccharide -binding protein, soluble CD163) | 10 hours after first intervention
plasma prolactin | 10 hours after first intervention
Plasma FSH | 10 hours after first intervention
Plasma LH | 10 hours after first intervention
plasma free testosterone | 10 hours after first intervention
plasma estradiol | 10 hours after first intervention
plasma keto-testosterone | 10 hours after first intervention
Homeostatic Model Assessment for Insulin Resistance | 10 hours after first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Rittig, Principal Investigator — University of Aarhus
Locations (1):
- Department of Diabetes and Hormone Diseases (DoH), Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rittig N, Christiansen Arlien-Soborg M, Svart MV, Thomsen HH, Kirkegaard K, Greve VH, Nielsen MM, Stochholm K, Ornstrup MJ, Gravholt CH. Ketone supplementation acutely lowers androgen and glucose levels in women with polycystic ovary syndrome: a randomized clinical trial. Eur J Endocrinol. 2025 May 30;192(6):717-727. doi: 10.1093/ejendo/lvaf106. PMID 40393075